CLINICAL TRIAL: NCT06331923
Title: Assessing the Effectiveness of Continuous Glucose Monitoring Compared with Conventional Monitoring in Enhancing Surgical Outcomes for Patients with Diabetes: a Multi-center, Parallel-arm, Randomized, Pragmatic Trial in China
Brief Title: Assessing the Effectiveness of Continuous Glucose Monitoring in Enhancing Surgical Outcomes for Patients with Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Peking University International Hospital (Other); Wang Jing Hospital (Other); ZhuHai Hospital (Other); Beijing Hospital (Other Government); Siyang County Hospital of Traditional Chinese Medicine (Unknown); Second Hospital of Shanxi Medical University (Other); Henan Provincial Chest Hospital (Other); Fuzhou First Hospital (Unknown); Pinggu Hospital of Beijing Traditional Chinese Medicine Hospital (Other); The First Affiliated Hospital of Anhui University of Chinese Medicine (Other); The First Affiliated Hospital of Zhengzhou University (Other); Mindong Hospital of Ningde (Unknown); The Fifth Hospital of Xiamen (Unknown); People's Hospital of Ningxia Hui Autonomous Region (Other); The First People's Hospital of Changzhou (Other); The Fifth hospital of Deyang (Unknown); Suzhou Municipal Hospital (Other); Tang-Du Hospital (Other); Yiyang Central Hospital (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); Peng Ding Shan Shi Zhong Yi Yi Yuan (Unknown); Yueyang Central Hospital (Other); The First People's Hospital of Lianyungang (Other); Haimen District Traditional Chinese Medicine Hospital (Unknown); The 910th Hospital (Unknown); The Second Affiliated Hospital of Zhejiang Chinese Medical University (Other); Beijing Tiantan Hospital (Other); Affiliated Hospital of Jiangsu University (Other); Liaocheng People's Hospital (Other); Beijing Chao Yang Hospital (Other); Jilin City Hospital of Chemical Industry (Unknown); Creen Hospital-465 (Unknown); Wuhan Central Hospital (Other); Air Force Military Medical University, China (Other); Shanghai Tong Ren Hospital (Other); Beijing Anzhen Hospital (Other); Emergency General Hospital (Other); Beijing Tongren Hospital (Other); Civil Aviation General Hospital (Other); Peking University Shougang Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Chinese PLA Central Hospital (Unknown)
Responsible Party: Principal Investigator, Zhifeng Gao, Deputy director, Department of Anesthesiology, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1305-0484
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Comprehensive Complication Index
Keywords: comprehensive complication index; continuous glucose monitoring; perioperative; prognosis
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGM group (Experimental): Participants who receive continuous glucose monitoring (CGM) during the perioperative period. Glucose monitoring should be continued until the 7th day after surgery or discharge.
  Interventions: Device: Continuous glucose monitoring (CGM) device
- Control group (No Intervention): Perioperative blood glucose monitoring was performed according to institutional treatment guidelines.Glucose monitoring should be continued until the 7th day after surgery or discharge.

INTERVENTIONS:
Device: Continuous glucose monitoring (CGM) device — Continuous glucose monitoring (CGM) will be prescribed by the attending physician for at least 6 hours before surgery. The supervising nurse will educate the patient and their family on the correct wearing and connection of the CGM device. The calibration frequency and interval of glucose monitoring devices before and after surgery should be determined according to institutional treatment guidelines and the requirements of the monitoring device used. Intraoperative glucose calibration should be done immediately upon entering the operating room, immediately after skin incision, every 2 hours after skin incision, and at the end of wound closure. Glucose monitoring should be continued until the 7th day after surgery or discharge.
  Arms: CGM group

SUMMARY:
The goal of this multi-center, pragmatic, randomized controlled trial is to assess the effectiveness of continuous glucose monitoring (CGM) compared with conventional monitoring in enhancing surgical outcomes for diabetic patients. The main questions it aims to answer are:

* To assess the effectiveness of CGM compared with conventional monitoring in reducing the comprehensive complication index (CCI) for patients with diabetes or impaired glucose tolerance (IGT) within 30 days after surgery.
* To analyze the impact of different age groups, types of surgery, preoperative levels of HbA1c, and preoperative 24h glycemic variations on the improvement of surgical outcomes under the CGM model.

Participants will receive CGM prescribed by the attending physician for at least 6 hours before surgery. Glucose monitoring should be continued until the 7th day after surgery or discharge.

The investigators will compare conventional monitoring group to see if CGM could reduce the CCIs for patients with diabetes or impaired glucose tolerance within 30 days after surgery.

DETAILED DESCRIPTION:
Abstract: Postoperative complications are important factors in reducing surgical quality and increasing healthcare costs. The CCI is an internationally recognized index to quantify postoperative complications. Patients with diabetes mellitus (DM) or IGT are more prone to developing dysglycemia during the perioperative period, which in turn leads to various types of complications and increased mortality, as evidenced by a significant increase in CCI. Our previous study confirmed that strict glucose management in the perioperative period can help reduce the incidence of postoperative complications such as surgical site infections (SSIs), but this strategy has not been replicated in the perioperative period due to the disadvantages of heavy and complex operations and the possible increased risk of concomitant hypoglycemia. CGM, with its advantages of portability, accuracy, real-time, and information-richness, has been used for precise glucose management in chronic diseases. A small number of prospective randomized controlled studies have previously demonstrated the existence of an improved effect of CGM on intraoperative glycemic management in major surgery. However, there are no real-world studies with large sample sizes to clarify the efficacy and safety of CGM in reducing CCI in patients with DM or IGT. This is where our research comes in. In this real-world study, we aim to clarify the role of perioperative CGM in improving both prognosis and efficacy of surgery.

This is an investigator-initiated, multi-center, pragmatic,1:1ratio randomized, parallel-group, controlled trial which consisted of a 1 to 3-day screening period, and a 7-day(at least 3-day) intervention period, with a final evaluation at day 30. A total of approximately 10168 patients (≥ 18 years of age) with DM or IGT undergoing elective surgeries (including major thoracoabdominal surgery [excluding cardiac surgery], open orthopedic surgery, or neurosurgery) will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized into two groups (CGM group versus C group) according to the 1:1 ratio after offering informed content.

Glucose monitoring models:

1. CGM group: A CGM prescription will be issued by the attending physician at least 6 hours before surgery. The primary nurse in charge will educate the participant and their family members on the proper wearing and connection of the CGM device. The calibration frequency and interval of preoperative and postoperative glucose monitoring devices will be determined based on institutional diagnostic and treatment guidelines and the requirements of the monitoring device used. Intraoperative glucose calibration will be performed immediately upon admission, immediately after surgical incision, every 2 hours after surgical incision, and at the completion of wound closure.
2. C group: Perioperative glucose monitoring will be conducted based on institutional diagnostic and treatment guidelines.
3. Glucose/blood glucose monitoring will be continued for both groups of patients until postoperative day 7 or discharge.

Perioperative glucose management:

1. Preoperatively: For elective surgery, preoperative fasting blood glucose/glucose ≤10 mmol/L and HbA1c≤7.0%. For emergency surgery, the decision whether the participant's current blood glucose level is acceptable for surgical treatment is based on institutional practice and the experience of the physician in charge.
2. Intraoperatively: Blood glucose level will be set at 4.5-10mmol/L. Participants in both groups will be given glucose to elevate blood glucose when blood glucose was found to be≤4.5 mmol/L, or insulin when blood glucose was found to be ≥10 mmol/L. Drug dosages and administration methods will follow the medical practice of the institution and the anaesthesiologist in charge. In the CGM group, if mean amplitude of glycemic excursions (MAGE) ≥3.9 mmol/L or largest amplitude of glycemic excursions (LAGE)≥4.4 mmol/L was found in the last 2 h, the dose or rate of glucose/insulin administration will be adjusted as appropriate.
3. Postoperatively: The target of blood glucose management in the early postoperative period is 4.5-7.8 mmol/L. According to the institutional practice and the supervising physician's experience, participants in both groups will be treated with glucose to elevate blood glucose when blood glucose was found to be ≤4.5 mmol/L, and will be treated with insulin to lower blood glucose when blood glucose was found to be ≥7.8 mmol/L.In the CGM group, if excessive blood glucose variability was found, including coefficient of variation (CV)≥36%, LAGE≥4.4 mmol/L, postprandial glucose excursions of three dinners (PPGE)≥2.2mmol/L, standard deviation of blood glucose (SDBG)≥2.0 mmol/L or time in range (TIR)≤70%, an endocrinologist will aid in adjusting the blood glucose management programme.

The primary objective is to observe the improvement of CGM on the surgical outcomes of participants with DM or IGT, including a reduction in the CCI, overall postoperative infection rate, major adverse cardiovascular events (MACE) rate, and shortened postoperative hospital stay within 30 days after surgery.

The study consists of 9 visits including the day of screening and randomization,1,2,3,4,5,6,7 and 30-day follow-up postoperatively.

Demographic information, symptoms and signs, laboratory test, auxiliary examinations, CCIs will be recorded during the program. The trial is anticipated to last from April 2024 to December 2025 with 10168 subjects recruited from 50 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese Good Clinical Practice standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by the ethics committee of Beijing Tsinghua Chang Gung Hospital and corresponding branch centers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged above 18 years;
2. Patients with diabetes mellitus or impaired glucose tolerance;
3. Expected major thoracic and abdominal surgery (except cardiac surgery; including endoscopic surgery and robotic surgery), open orthopedic surgery, neurosurgery;
4. Volunteered for this study and written informed consent.

Exclusion Criteria:

1. The patient refused;
2. The time between wearing CGM sensor and surgical skin incision cannot meet 6 hours or more;
3. Expected monitoring time less than 72 hours in CGM group;
4. Patients had comorbidities that affected the evaluation of endpoints;
5. The attending physician thought that the patient had inappropriate indications for enrollment;
6. Participants were involved in other studies that interfered with the evaluation of the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10168 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive complication index | At 30-day follow-up
  The investigators will use the online tool（www.assesssurgery.com）to calculate every participant's cumulative comprehensive complication index (CCI) at 30-day follow-up. CCI is a validated prognostic assessment tool that calculates the total score of all complications weighted by severity, ranging from 0 (no complications) to 100 (death) for each patient. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Postoperative complications | At 1-7 day postoperatively and 30-day follow-up
  Postoperative complications will be diagnosed abased on signs, symptoms, laboratory and auxiliary examinations.
Mortality | At 30-day follow-up
  Mortality will be expressed by the number and percentage of occurrences.
Perioperative glucose level | Perioperative glucose level will be monitored from the day of the enrollment to 7 days (at least 3 days) postoperatively.
  CGM group: using CGM device; Control group: using conventional glucose monitoring, such as arterial blood gas, biochemistry examinations.
The length of the stay in the intensive care unit | At 30-day follow-up
  The investigators will search the medical archives of participants.
The overall hospitalization cost | At 30-day follow-up
  The investigators will search the medical archives of participants.

OTHER OUTCOMES:
Incidence of postoperative infection | Within 30 days after surgery
  Postoperative infection will be expressed by the number and percentage of occurrences.
Incidence of major adverse cardiovascular event (MACE) | Within 30 days after surgery
  MACE includes cardiovascular death, myocardial infarction, stroke, urgent revascularization, hospitalization for heart failure, recurrent angina, and severe arrhythmias. MACE rate will be expressed by the number and percentage of occurrences.
Incidence of stroke | Within 30 days after surgery
  Stroke will be assessed through clinical manifestations, auxiliary examinations, and relevant scale (National Institute of Health Stroke Scale [NIHSS]). NIHSS scale rangs from 0 to 42 for each patient. Higher values represent a worse outcome. Stroke rate will be expressed by the number and percentage of occurrences.
The length of hospital stay | At 30-day follow-up
  The investigators will search the medical archives of participants.
Incidence of delirium | Within 30 days after surgery
  Delirium will be assessed through clinical manifestations, auxiliary examinations, and Confusion Assessment Method (CAM). Delirium will be expressed by the number and percentage of occurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Yao, Principal Investigator — Peking University International Hospital; Hui Q Xu, Principal Investigator — Wangjing Hospital, China Academy of Chinese Medical Sciences; Yan Liu, Principal Investigator — ZhuHai Hospital; Qi Pan, Principal Investigator — Beijing Hospital; Jian H Jia, Principal Investigator — Siyang County Hospital of Traditional Chinese Medicine; Yi K Zhu, Principal Investigator — Second Hospital of Shanxi Medical University; Ke F Shi, Principal Investigator — Henan Provincial Chest Hospital; Fang F Zhang, Principal Investigator — Fuzhou First Hospital; Xiu Zh Wang, Principal Investigator — Pinggu District Hospital of Traditional Chinese Medicine; Feng Hong, Principal Investigator — The First Affiliated Hospital of Anhui University of Chinese Medicine; Ying J Hao, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Yi Q Cai, Principal Investigator — Mindong Hospital of Ningde; Lin Shen, Principal Investigator — Heze Hospital of Traditional Chinese Medicine; Jin L Liang, Principal Investigator — The Fifth Hospital of Xiamen; Zhen Wang, Principal Investigator — People's Hospital of Ningxia Hui Autonomous Region; Hong W Ye, Principal Investigator — The First People's Hospital of Changzhou; Qin Wang, Principal Investigator — The Fifth hospital of Deyang; Jian P Qiu, Principal Investigator — Suzhou Municipal Hospital; Bo Liao, Principal Investigator — Tang-Du Hospital; Xin J Liu, Principal Investigator — Yiyang Central Hospital; Guo Sh Gu, Principal Investigator — Anhui No.2 Provincial People's Hospital; Li Quan, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Li R Ma, Principal Investigator — Peng Ding Shan Shi Zhong Yi Yi Yuan; Zhi B Zhao, Principal Investigator — The First People's Hospital of Lianyungang; Xin Lu, Principal Investigator — Haimen District Traditional Chinese Medicine Hospital; Feng Zhou, Principal Investigator — Yueyang Central Hospital; Xiao D Yin, Principal Investigator — Zhe Cheng TCM Hospital; Li T Zhang, Principal Investigator — The 910th Hospital; Yu Zh He, Principal Investigator — The Second Affiliated Hospital of Zhejiang Chinese Medical University; Xiao M Zhang, Principal Investigator — The first People's Hospital of Zhengzhou; Yu H Jiang, Principal Investigator — Beijing Tiantan Hospital; Peng Jiang, Principal Investigator — Affiliated Hospital of Jiangsu University; Xiao Y Li, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Zhi H Liu, Principal Investigator — Liaocheng People's Hospital Zhiheng Liu; Jin C Yang, Principal Investigator — Beijing Chao Yang Hospital; Xue L Zhu, Principal Investigator — The People's Hospital of Nanchuan, Chongqing; Wen T Si, Principal Investigator — Zhengzhou Orthopaedic Hospital; Lei Ning, Principal Investigator — Jilin City Hospital of Chemical Industry; Li H Su, Principal Investigator — Creen Hospital-465; Zhong J Wang, Principal Investigator — Wuhan Central Hospital; Li P Ma, Principal Investigator — Beijing Anzhen Hospital; Yu H Xu, Principal Investigator — Air Force Military Medical University, China; Jiang M Yu, Principal Investigator — Tong Ren hospital Shanghai Jiao Tong university school of medicine; Qing H Cheng, Principal Investigator — Emergency General Hospital; Hui J Wang, Principal Investigator — Beijing Tongren Hospital, CMU; Jun Wu, Principal Investigator — Heilongjiang provincial hospital; Jun T Duan, Principal Investigator — Civil Aviation General Hospital; Zheng G Guo, Principal Investigator — Peking University Shougang Hospital; Xin Kuang, Principal Investigator — The People's Hospital of Longhua, Shenzhen; Chang J Yu, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Feng Liang, Principal Investigator — Chinese PLA Central Hospital
Locations (1):
- Zhifeng Gao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data are not publicly available due to containing information that could compromise the privacy of research participants. The data that support the findings of this study are available on request from the corresponding author.

REFERENCES:
- [Derived] Duan Y, Ding L, Gao Z, Wang Y, Cao H, Zhang H, Yao L. Assessing the effectiveness of continuous glucose monitoring compared with conventional monitoring in enhancing surgical outcomes for patients with diabetes: protocol for a multicentre, parallel-arm, randomised, pragmatic trial in China. BMJ Open. 2025 Feb 18;15(2):e090664. doi: 10.1136/bmjopen-2024-090664. PMID 39965943